CLINICAL TRIAL: NCT07039227
Title: Evaluation of the Prognostic Value of Immature Platelet Fraction in Septic Patients Admitted to Critical Care
Brief Title: Evaluation of the Prognostic Value of Immature Platelet Fraction
Acronym: IPSIS
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/314/OB; N° IDRCB : 2022-A02612-41 (Other: ANSM)
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-05

CONDITIONS: Septic Shock
Keywords: coagulation; highlighting of biomarkers
MeSH Terms: conditions — Shock, Septic; Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Years
Biospecimen Retention: Samples Without DNA — At each patient follow-up time (At enrollment visit, 1-day visit, 3-day visit, 7-day visit), 4 tubes of 4 mL of blood will be collected (a total of 16 mL): 2 EDTA tubes for research, 1 citrated tube and one dry tube.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis Group: Patient admitted for sepsis in critical care
- Inflammatory control group: Patient admitted for an anesthesia consultation for cardiac surgery under extracorporeal circulation

SUMMARY:
Sepsis is a public health issue responsible for six million deaths worldwide each year. It is one of the leading causes of admission and morbidity and mortality in critical care. Its most severe form, septic shock, is responsible for a picture of multiple organ failure syndrome with a high mortality rate estimated at 38%. It appears important to identify routinely available and low-cost biomarkers to identify patients at risk of adverse outcomes.

DETAILED DESCRIPTION:
In the pathophysiology of host defense against infection, coagulation plays a major role. In the most severe forms of sepsis, there is an activation of coagulation, particularly platelets, which can cause an alteration of microcirculation and contribute to organ failure. This mechanism is called thromboinflammation. The appearance of thrombocytopenia in sepsis is a risk factor for severity and intrahospital mortality. Immature (or reticulated) platelets are young platelets that have just been released by the bone marrow. They are more prothrombotic and hyperactive than more mature platelets. They are a good marker of thrombopoiesis and platelet renewal, and can be easily obtained routinely on a complete blood count. Several studies show that the immature platelet count and/or fraction (IPF) could be a useful tool for predicting the development of sepsis and its severity. It appears interesting to study these IPFs in patients with sepsis to identify them and implement more aggressive therapies to prevent adverse outcomes in these patients. To distinguish between sepsis and inflammation and validate this marker, it will be compared to an inflammatory group using patients who underwent cardiopulmonary bypass as part of cardiac surgery.

The main objective of this study is to investigate the potential impact of the immature platelet fraction on the prognosis at day 28 of patients admitted to critical care for sepsis or septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient admitted to critical care for sepsis defined by a SOFA score > or = 2 or an increase of at least 2 points if there was organ dysfunction pre-existing to the infection.
* For the inflammatory control group, we will include adult patients who have required extracorporeal circulation for more than 1 hour for cardiac surgery.
* Patients who have read and understood the information letter and do not object to participating in the study
* Patients affiliated with a social security scheme
* Exclusion Criteria:
* Patient refusal
* Pregnant, parturient, or breastfeeding woman
* Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection/guardianship or curatorship
* Person who does not understand or speak French
* Moribund
* Febrile aplasia
* Hematological diseases
* Decompensated cirrhosis
* Ongoing chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to critical care for sepsis or septic shock
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the impact of the immature platelet fraction of patients admitted to intensive care for sepsis or septic shock on their prognosis at day 28. | Days 28
  Measurement of the fraction of immature platelets at admission in patients with sepsis or septic shock defined by the composite criterion calculated on the occurrence of death at 28 days of follow-up
Evaluation of the impact of the immature platelet fraction of patients admitted to intensive care for sepsis or septic shock on their prognosis at day 28. | Days 28
  Measurement of the fraction of immature platelets at admission in patients with sepsis or septic shock defined by the composite criterion calculated on the occurrence of organ failure: implementation of extrarenal purification and/or renal failure KDIGO 3 and/or moderate to severe acute respiratory distress syndrome and/or intense vasoplegic septic shock with noradrenaline > 0.25 µg/kg/min or vasopressin > 0.02 IU/h and/or myocardial dysfunction with venous oxygen saturation < 60 or a cardiac index < 2.2 l/min/m2 and/or occurrence of disseminated intravascular coagulation (DIC)

SECONDARY OUTCOMES:
To assess the impact of the immature platelet fraction on the occurrence of thrombocytopenia | days 28
  Occurrence of thrombocytopenia defined by a fall > or = to 30% of its baseline value or a platelet count < less than 150,000 G/L
Assess the impact of the immature platelet fraction on the progression to disseminated vascular coagulopathy | Days 28
  Demonstration of disseminated intravascular coagulation (DIC)
Evaluation of the impact of the immature platelet fraction on the occurrence of thromboembolic events | Days 28
  Evidence of the onset of thromboembolic venous disease
Assessment of the occurrence of multiple organ failure syndrome | Days 28
  Evidence of a multi-organ failure syndrome defined by the occurrence of at least 2 organ failures
Assessment of the occurrence of recourse to mechanical ventilation | Days 28
  Highlighting the use of mechanical ventilation
Assessment of mortality in intensive care, in hospital and on D28 | At enrollment visit, day 1, days 3, days 7 and Days 28
  Determination of Mortality in intensive care, in hospital and on D28

CONTACTS AND LOCATIONS:
Overall Officials: Perrine PL LEPRETRE, Doctor, Study Director — University Rouen Hospital
Locations (1):
- University Rouen Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No
The data provided will be the property of the sponsor and will be used solely for its own research activities.